CLINICAL TRIAL: NCT02919735
Title: A Randomized, Double Blind, Single Center, Controlled Study to Compare the Efficacy, Safety and Tolerability of CG 428 Cutaneous Solution With Placebo on Alopecia in Cancer Female Patients Under Chemotherapy
Brief Title: Efficacy, Safety and Tolerability of CG428 Cutaneous Solution on Chemotherapy Induced Alopecia; Controlled Study (ELAN)
Acronym: ELAN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Legacy Healthcare SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: ELAN
Record Dates: First submitted 2016-09-18; First posted 2016-09-29 (Estimated); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Alopecia
Keywords: Alopecia; Hair; Chemotherapy; Cancer
MeSH Terms: conditions — Alopecia; Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CG 428 cutaneous solution (Experimental): Herbal Medicinal Product, topical use by spray on the scalp
  Interventions: Drug: CG 428 cutaneous solution
- Placebo cutaneous solution (Placebo Comparator): Placebo, topical use by spray on the scalp
  Interventions: Drug: Placebo cutaneous solution

INTERVENTIONS:
Drug: CG 428 cutaneous solution — The patient will spray treatment 10 times directly to the scalp area, with the cannula, and then gently massage the whole scalp with fingertips, twice a day, spaced out by minimum 4 hours
  Arms: CG 428 cutaneous solution
Drug: Placebo cutaneous solution — The patient will spray treatment 10 times directly to the scalp area, with the cannula, and then gently massage the whole scalp with fingertips, twice a day, spaced out by minimum 4 hours
  Arms: Placebo cutaneous solution

SUMMARY:
Phase II clinical trial

DETAILED DESCRIPTION:
The aim of this trial is to compare the degree of efficacy, safety and tolerability of CG 428 cutaneous solution versus placebo on prevention of chemotherapy induced alopecia (CIA) in female patients with metastatic cancer treated with selected regimens inducing alopecia.

ELIGIBILITY:
Inclusion Criteria:

* Adult female, age ≥ 18 years.
* Patient with cancer, requiring one of the following pre-specified chemotherapy regimen according to local guidelines: weekly paclitaxel, weekly docetaxel, eribuline or associationof weekly paclitaxel/docetaxel with carboplatine (association of targeted therapies not influencing significantly the risk of alopecia is allowed, i.e. trastuzumab, pertuzumab or bevacizumab).
* Healthy hair (no current alopecia or scalp disease treatment).
* Life expectancy ≥ 6 months.
* Able to use the study treatment in compliance with the protocol.
* Physical and psychological ability to participate.
* Negative serum pregnancy test within 14 days prior to randomization in premenopausal women with childbearing potential.
* Patients must agree to not shave their head (minimum ≥ 1 cm).
* Signed and dated informed consent.

Exclusion Criteria:

* Other ongoing anti-neoplastic therapy or other investigational drug with potential effect on hair growth.
* Patients treated with proteasome inhibitors, i.e. bortezomib.
* Prior radiotherapy to the scalp with residual alopecia.
* Known allergy or hypersensitivity to some components of CG 428 cutaneous solution (including allium cepa (onion), citrus, caffeine, theobromine).
* Pre-existing alopecia or significant scalp disease, which may alter study treatment administration or absorption.
* Concomitant use of cold cap or any other anti-hair loss treatment.
* Hair transplants.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Rate of hair loss at different time points based of on Olsen's Visual Analog Scale (OVAS) and using the Severity of Alopecia Tool score (SALT score) | Every 3 to 8 weeks (variable). The following investigations will be performed every 3 to 4 weeks during the study treatment
  Physical examination of the scalp: skin AEs, hair status (alopecia graded according to CTCAE v.4.03.)

SECONDARY OUTCOMES:
Rate of grade 2 alopecia according to CTCAE v. 4.03. | Every 3 weeks for 24 weeks.
  CTCAE v. 4.03 : Common Toxicity Criteria for Adverse Event (skin toxicity)
Time to reach grade 2 alopecia during chemotherapyaccording to CTCAE v. 4.03. . | Every 3 weeks for 24 weeks.
  CTCAE v. 4.03 : Common Toxicity Criteria for Adverse Event (skin toxicity)
Time to recover to grade 1 and grade 0 according to CTCAE v. 4.03 after the last dose of the selected chemotherapy | Every 3 weeks for 24 weeks.
  CTCAE v. 4.03 : Common Toxicity Criteria for Adverse Event (skin toxicity)
Percent of hair loss according to OVAS (Olsen's visual analog scale) at different time points after the end of the chemotherapy. | Every 3 to 8 weeks (variable). The following investigations will be performed every 3 to 4 weeks during the study treatment
  Olsen's visual analog scale : visual aid for estimating percentage scalp hair loss.
Adverse events based on the CTCAE 4.03. | Every 3 to 8 weeks (variable). The following investigations will be performed every 3 to 4 weeks during the study treatment
Patient's subjective assessment through questionnaire | Every 3 weeks for 24 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Khalil KZ ZAMAN, Principal Investigator — Department Oncology - CHUV, 1011 Lausanne - CH
Locations (1):
- CHUV Lausanne, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: Yes